CLINICAL TRIAL: NCT04268316
Title: Virtual Reality Behavioral Activation: An Intervention for Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Margot Paul, Principle Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 53483
Record Dates: First submitted 2020-02-05; First posted 2020-02-13 (Actual); Results first posted 2021-05-10 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Major Depressive Disorder; MDD; Depression
Keywords: virtual reality; behavioral activation; depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either BA in VR, BA in real-life, or a waitlist control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (3):
- Virtual Reality Behavioral Activation (Experimental): Participants randomized to this arm will perform all of their behavioral activation in virtual reality. Participants will meet with the clinician once a week for three weeks (4 sessions). In between weekly therapy sessions, participants will pick four pleasurable activities to enjoy in virtual reality.
  Interventions: Device: Virtual Reality Behavioral Activation
- Behavioral Activation in real-life (Active Comparator): Participants randomized to this arm will perform all of their behavioral activation in real life. Participants will meet with the clinician once a week for three weeks (4 sessions). In between weekly therapy sessions, participants will pick four pleasurable or mastery activities to perform in real life.
  Interventions: Behavioral: Behavioral Activation in real-life
- Waitlist Control (No Intervention): Participants randomized to this arm will not receive any type of intervention and will be asked to complete the PHQ-9 once a week for three weeks (4 sessions) to track symptoms. Participants will be offered to engage in behavioral activation in real life or with virtual reality when the four weeks are complete. Their data will only be used from the time they were on the waitlist.

INTERVENTIONS:
Device: Virtual Reality Behavioral Activation — Participants will choose four "activities" to complete in virtual reality over the course of the week. These activities are video 360 and range from viewing animals, to viewing nature scenes, to traveling to a different location in the world, to viewing adrenaline-pumping activities.
  Arms: Virtual Reality Behavioral Activation
Behavioral: Behavioral Activation in real-life — Participants will choose four pleasurable and/or mastery activities to complete over the course of the week in real life.
  Arms: Behavioral Activation in real-life

SUMMARY:
The primary purpose of this study is to test the safety and feasibility of virtual reality (VR) technology in the use of behavioral activation (BA) as a treatment for major depressive disorder (MDD). The secondary purpose of this study is to examine whether any evidence of clinical efficacy exists for VR delivered BA.

DETAILED DESCRIPTION:
This is a treatment development trial. Participants will be randomly assigned to BA in VR, BA in real-life, or a waitlist control group. The former two groups will follow a BA protocol developed for primary care settings over a four-week treatment period. This study is taking place over Zoom, due to COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Patient must meet DSM V criteria for MDD
* Patient must be at least 18 years of age
* Patient must be English speaking

Exclusion Criteria:

* Substance Use Disorders in past year
* Any psychosis or bipolar I disorder
* Any seizure in the last 6 months or untreated epilepsy
* Current nonsuicidal self-injury or parasuicidal behavior
* Current suicidal urges and intent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Bullock, MD, Study Director — Stanford University; Margot Paul, MS, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No
No current plan to share data.

REFERENCES:
- [Result] Paul M, Bullock K, Bailenson J. Virtual Reality Behavioral Activation as an Intervention for Major Depressive Disorder: Case Report. JMIR Ment Health. 2020 Nov 3;7(11):e24331. doi: 10.2196/24331. PMID 33031046
- [Derived] Paul M, Bullock K, Bailenson J. Virtual Reality Behavioral Activation for Adults With Major Depressive Disorder: Feasibility Randomized Controlled Trial. JMIR Ment Health. 2022 May 6;9(5):e35526. doi: 10.2196/35526. PMID 35404830

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 20 participants signed consent, but only 13 participants were randomized to a study arm.
Groups:
- Virtual Reality Behavioral Activation: Participants engage in VR activities over the week for three weeks.
- Behavioral Activation in Real-life: Participants engage in real life pleasurable activities over the week for three weeks.
- Waitlist Control: Participants answer the PHQ-9 weekly for four sessions.
Period: Overall Study
Arm/Group | Virtual Reality Behavioral Activation | Behavioral Activation in Real-life | Waitlist Control
Started | 5 | 4 | 4
Completed | 3 | 3 | 4
Not Completed | 2 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Virtual Reality Behavioral Activation | Behavioral Activation in Real-life | Waitlist Control | Total
Number analyzed (Participants) | 5 | 4 | 4 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.6 (9.2) | 46 (15.7) | 29.5 (5.2) | 35.4 (12.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  male | 1 | 3 | 1 | 5
  female | 4 | 1 | 2 | 7
  non-binary/third gender | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic Caucasian | 3 | 3 | 1 | 7
  Chinese | 1 | 1 | 0 | 2
  Indian | 1 | 0 | 0 | 1
  African American | 0 | 0 | 1 | 1
  Mexican | 0 | 0 | 1 | 1
  Hispanic/Latino | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 4 | 4 | 13
Patient Health Questionnaire-9 (PHQ-9) [Mean (Standard Deviation); unit: score on a scale] — Total Score Depression Severity
  * 0 Lack of depression symptoms
  * 1-4 Minimal depression
  * 5-9 Mild depression
  * 10-14 Moderate depression
  * 15-19 Moderately severe depression
  * 20-27 Severe depression Population: Participants that completed the protocol are included in the analysis.
  score on a scale
    number analyzed (Participants) | 3 | 3 | 4 | 10
    (all) | 14.3 (5.7) | 15.3 (4.9) | 14 (4.1) | 14.5 (4.3)

OUTCOME MEASURES:

1. Primary Outcome: Participant's Desire to Continue Using VR After the Study Ends
Description: This outcome was measured using the "Intention to use Technology " questions of the Technology Acceptance Model questionnaire. These are questions 11, 12, and 13 and allow participants the option of circling Strongly Disagree (0), Disagree (1), Neutral (2), Agree (3), or Strongly Agree (4). With 3 questions, the total range was 0-12 (higher scores indicate greater acceptance).
Time Frame: Assessed at the end of week 3, after session 4
Population: This outcome measure was assessed in the Virtual Reality Behavioral Activation group only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality Behavioral Activation
Number analyzed (Participants) | 5
score on a scale | 9.54 (2.5)

2. Primary Outcome: Number of Participants Who Dropped Out of Each Study Arm
Description: Participant treatment dropout was compared across each study arm. This was reported as the count of participants who discontinued the study for any reason.
Time Frame: 3-weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Reality Behavioral Activation | Behavioral Activation in Real-life | Waitlist Control
Number analyzed (Participants) | 5 | 4 | 4
Participants | 2 | 1 | 0

3. Primary Outcome: Participant's Satisfaction With the VR-BA Treatment
Description: This outcome was measured using the "Attitudes Toward Use " questions of the Technology Acceptance Model questionnaire. These are questions 7, 8, 9, and 10 and allow participants the option of circling Strongly Disagree (0), Disagree (1), Neutral (2), Agree (3), or Strongly Agree (4). With 4 questions, the total range was 0-16 (higher scores indicate greater acceptance).
Time Frame: Assessed at the end of week 3, after session 4
Population: This outcome measure was assessed in the Virtual Reality Behavioral Activation group only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality Behavioral Activation
Number analyzed (Participants) | 5
score on a scale | 12.5 (3.5)

4. Primary Outcome: Participant's Use of the VR Headset
Description: This was measured by noting the amount of times the VR headset is used during the 3-week study period.
Time Frame: Assessed at the end of week 3, after session 4
Population: This outcome measure was assessed in the Virtual Reality Behavioral Activation group of protocol completers only.
Measure: Mean (Standard Deviation); unit: times used
Arm/Group | Virtual Reality Behavioral Activation
Number analyzed (Participants) | 3
times used | 21.7 (11)

5. Primary Outcome: Participant's Acceptance of VR-BA Treatment
Description: This was measured using the overall Technology Acceptance Model questionnaire, which encompasses 13 questions and allows participants the option of circling Strongly Disagree (0), Disagree (1), Neutral (2), Agree (3), or Strongly Agree (4), yielding a range of 0-52 (higher scores indicate greater acceptance).
Time Frame: Assessed at the end of week 3, after session 4
Population: This outcome measure was assessed in the Virtual Reality Behavioral Activation group only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality Behavioral Activation
Number analyzed (Participants) | 5
score on a scale | 42.4 (8.4)

6. Primary Outcome: How Well Can Participants Tolerate the VR-BA Treatment?
Description: This was determined by the Simulator Sickness Questionnaire, which names 16 adverse symptoms and asks participants to circle as compared to baseline: No more than usual (0), Slightly more than usual (1), Moderately more than usual (2), or Severely more than usual (3), yielding a range of 0-48 (lower scores indicate greater tolerability).
Time Frame: Assessed at the end of week 3, after session 4
Population: This outcome measure was assessed in the Virtual Reality Behavioral Activation group only.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Virtual Reality Behavioral Activation
Number analyzed (Participants) | 5
score on a scale | 2.9 [0.4 to 8.7]

7. Primary Outcome: How Present Did Individuals in the VR-BA Treatment Feel?
Description: This was measured using the Presence Questionnaire, which asks three questions and asks the participants to circle either Not at all (0), Slightly (1), Moderately (2), Strongly (3), or Very Strongly (4), yielding a range of 0-12 (higher scores indicate greater presence).
Time Frame: Assessed at the end of week 3, after session 4
Population: This outcome measure was assessed in the Virtual Reality Behavioral Activation group only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality Behavioral Activation
Number analyzed (Participants) | 5
score on a scale | 7.1 (2.8)

8. Secondary Outcome: Change in Depression Scores on the PHQ-9 From Baseline to Session 4, Compared Across Three Study Arms
Description: How participants' depression scores on the Patient Health Questionnaire (PHQ-9) change over time using VR-BA compared to BA in real life and a waitlist control. The PHQ-9 is a 9-question screener with a score range of 0-29, with 29 indicating the most severe depression and 0 indicating a lack of depression symptoms. The greater the change over time, the greater the symptom reduction.
Time Frame: Assessed at baseline and session 4.
Population: Protocol Completers
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Virtual Reality Behavioral Activation | Behavioral Activation in Real-life | Waitlist Control
Number analyzed (Participants) | 3 | 3 | 4
score on a scale | 5.7 [2 to 12] | 3 [2 to 5] | .25 [-5 to 3]

ADVERSE EVENTS:
Time Frame: 3-weeks
Arm/Group | Virtual Reality Behavioral Activation | Behavioral Activation in Real-life | Waitlist Control
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/4

LIMITATIONS AND CAVEATS:
This study did not enroll to its planned sample size of 30.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-02-25): https://cdn.clinicaltrials.gov/large-docs/16/NCT04268316/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-13): https://cdn.clinicaltrials.gov/large-docs/16/NCT04268316/SAP_001.pdf